CLINICAL TRIAL: NCT02561130
Title: Remission Evaluation of a Metabolic Intervention in Type 2 Diabetes With Forxiga
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT-Dapa
Record Dates: First submitted 2015-09-16; First posted 2015-09-25 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Insulin; Glargine; Metformin; Forxiga; Diet; Exercise; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Motor Activity | interventions — Insulin Glargine; Metformin; dapagliflozin; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Drug: insulin glargine - sc injection; Drug: metformin, oral administration; Drug: forxiga, oral administration; Behavioral: lifestyle therapy, diet and exercise
  Interventions: Drug: insulin glargine; Drug: metformin; Drug: Forxiga; Behavioral: Lifestyle therapy
- Standard Care (No Intervention): Standard glycemic care as informed by the current clinical practice guidelines

INTERVENTIONS:
Drug: insulin glargine — Dose is titrated to achieve fasting normoglycemia
  Other Names: Lantus
  Arms: Intervention
Drug: metformin — Dose is titrated to 1 g bid or maximal tolerated dose
  Arms: Intervention
Drug: Forxiga — Dose is titrated to 10 mg po daily or maximal tolerated dose
  Other Names: dapagliflozin
  Arms: Intervention
Behavioral: Lifestyle therapy — Lifestyle intervention includes individualized dietary and exercise advice and frequent visits for goal reinforcement, behavior modification and problem-solving
  Other Names: diet and exercise
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine whether in patients with early type 2 diabetes, a short-term intensive metabolic intervention comprising Forxiga, metformin, basal insulin glargine and lifestyle approaches will be superior to standard diabetes therapy in achieving sustained diabetes remission.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized controlled trial in 152 patients with recently-diagnosed T2DM. Participants will be randomized to 2 treatment groups: (a) a 12-week course of treatment with Forxiga, metformin, insulin glargine and lifestyle therapy, and (b) standard diabetes therapy, and followed for a total of 64 weeks (1 year and 3 months). In all participants with HbA1C<7.3% at the 12 week visit, glucose-lowering medications will be discontinued and participants will be encouraged to continue with lifestyle modifications and regular glucose monitoring. Participants with HbA1C ≥ 7.3% at this visit or who experience hyperglycemia relapse after stopping drugs will receive standard glycemic management as informed by the current Canadian Diabetes Association clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. men and women 30-80 years of age inclusive;
2. type 2 diabetes mellitus diagnosed by a physician within 8 years prior to patient enrollment;
3. anti-diabetic drug regimen (either drug or dose of drug) unchanged during 8 weeks prior to screening and randomization;
4. HbA1C 6.5-9.5% inclusive on no hypoglycemic agents or HbA1C ≤ 8.0% on up to 2 glucose-lowering agents;
5. body mass index ≥ 23 kg/m2;
6. ability and willingness to perform self-monitoring of capillary blood glucose (SMBG);
7. ability and willingness to self-inject insulin;
8. provision of informed consent.

Exclusion Criteria:

1. current use of insulin therapy;
2. history of hypoglycemia unawareness, or severe hypoglycemia requiring assistance;
3. history of end-stage renal disease or renal dysfunction as evidenced by eGFR<60 mL/min/1.73 m2 by MDRD formula;
4. history of lactic acidosis or diabetic ketoacidosis;
5. active liver disease or elevated alanine transferase (ALT) levels ≥ 2.5 times upper limit of normal at the time of enrollment;
6. history of bladder cancer or undiagnosed hematuria;
7. history of breast cancer;
8. history of polycythemia;
9. evidence of volume depletion or hypotension (systolic blood pressure < 90 mmHg);
10. systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg;
11. diagnosed cardiovascular disease (unless cleared for a moderate intensity exercise program by a specialist) including:

    1. any history of acute coronary syndrome, hospitalization for unstable angina, myocardial infarction, or revascularization with coronary artery bypass grafting or percutaneous coronary intervention;
    2. other evidence of coronary artery disease;
    3. peripheral vascular disease, valvular heart disease, cardiomyopathy, aortic dissection, tachyarrhythmias, bradyarrhythmias, prior stroke or TIA;
    4. prior hospitalization for heart failure; or
    5. ECG findings concerning for ischemic heart disease (i.e. pathological Q-waves, ST-segment-T-wave abnormalities in contiguous leads, left anterior hemiblock, left bundle branch block, second or third degree atrioventricular block).
12. dependence on oxygen;
13. history of any disease requiring frequent intermittent or continuous systemic glucocorticoid treatment;
14. history of bariatric surgery, or planned bariatric surgery in the next 1.5 years;
15. history of any major illness with a life expectancy of < 3 years;
16. history of injury or any other condition that significantly limits participant's ability to achieve moderate levels of physical activity;
17. any history of excessive alcohol intake, acute or chronic;
18. currently pregnant, or breastfeeding, or not using a reliable method of birth control for the duration of the trial in all females with childbearing potential; reliable methods of birth control include oral contraceptive (birth control pill), hormonal injection, implant, patch, or vaginal ring, intrauterine device, barrier method (condom and spermicide), tubal ligation, partner vasectomy or abstinence;
19. known hypersensitivity to metformin, Forxiga, or insulin glargine.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia McInnes, MD, Principal Investigator — McMaster University; Hertzel C Gerstein, MD, Study Chair — Hamilton Health Sciences Corporation
Locations (7):
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Health Science Centre, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Western University, London, Ontario
  - LMC, Toronto, Ontario
  - St. Michaels's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] McInnes N, Hall S, Sultan F, Aronson R, Hramiak I, Harris S, Sigal RJ, Woo V, Liu YY, Gerstein HC. Remission of Type 2 Diabetes Following a Short-term Intervention With Insulin Glargine, Metformin, and Dapagliflozin. J Clin Endocrinol Metab. 2020 Aug 1;105(8):dgaa248. doi: 10.1210/clinem/dgaa248. PMID 32403130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Standard Care
Started | 77 | 77
Completed | 76 | 76
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard Care | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.0) | 56.7 (9.6) | 56.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 50 | 50 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 64 | 61 | 125
  Non-Caucasian | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  Canada | 77 | 77 | 154
Duration of diabetes [Mean (Standard Deviation); unit: months] | 37.7 (26.7) | 35.8 (27.8) | 36.8 (27.2)
Glycated hemoglobin (HbA1C) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — Expressed in Diabetes Control and Complications Trial (DCCT) units
  percentage of glycated hemoglobin | 6.7 (0.6) | 6.7 (0.7) | 6.7 (0.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (5.8) | 32.5 (6.0) | 32.9 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Drug-free Diabetes Remission in the Experimental Group Compared to the Control Group
Description: Drug-free diabetes remission is defined as HbA1C < 6.5 % off glucose-lowering agents for at least 12 weeks.
Time Frame: 24 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 19 | 13

2. Secondary Outcome: Number of Participants Achieving Drug-free Diabetes Remission
Description: Drug-free diabetes remission is defined as HbA1C < 6.5 % off glucose-lowering agents for at least 12 weeks.
Time Frame: 64 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 11 | 6

3. Secondary Outcome: Number of Participants Achieving Drug-free HbA1C < 6.0%
Description: Drug-free complete diabetes remission is defined as HbA1C < 6.0 % off glucose-lowering agents for at least 12 weeks.
Time Frame: 24 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 6 | 6

4. Secondary Outcome: Number of Participants Achieving Diabetes Relapse Without Overt Hyperglycemia Off Diabetes Drugs
Description: Diabetes relapse without overt hyperglycemia is defined as HbA1C 6.5-6.9% off glucose-lowering agents for at least 12 weeks.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 20 | 9

5. Secondary Outcome: Glycated Hemoglobin (HbA1C)
Description: Expressed in Diabetes Control and Complications Trial (DCCT) units
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 66
percentage of glycated hemoglobin | 5.9 (0.4) | 6.6 (0.7)

6. Secondary Outcome: Number of Participants With Non-severe Symptomatic Hypoglycemic Episodes
Description: Symptomatic hypoglycemic episode is defined as an event with clinical symptoms consistent with hypoglycemia.
Time Frame: During 64 weeks of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 34 | 15

7. Secondary Outcome: Percentage of Weight Loss From Baseline
Description: (Weight at randomization - weight at 12 weeks)/(weight at randomization)
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 76 | 64
percentage of weight loss | 2.9 (3.2) | 1.0 (2.5)

8. Secondary Outcome: Change in Waist Circumference From Baseline
Description: (Waist circumference at 12 weeks - waist circumference at randomization)
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 76 | 64
cm | -3.0 (4.1) | -1.3 (3.3)

9. Secondary Outcome: Number of Participants With Severe Hypoglycemic Episodes
Description: Severe hypoglycemic episode is defined as an event with clinical symptoms consistent with hypoglycemia in which the participant required the assistance of another person, and one of the following: (i) the event was associated with a documented self-measured or laboratory plasma glucose level </= 2.0 mmol/L or (ii) the event was associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration.
Time Frame: During 64 weeks of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 77 | 77
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 64 weeks
Arm/Group | Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 3/77 | 0/77
Other Adverse Events (participants affected / at risk) | 12/77 | 10/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=77) | Standard Care (N=77)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Resection of liver metastases from colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=77) | Standard Care (N=77)
Genitourinary infection (Infections and infestations) | 4 (5) | 1 (1)
Other infections (Infections and infestations) | 0 (0) | 3 (3)
Abscess drainage (Infections and infestations) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Abdominal pain (General disorders) | 3 (3) | 0 (0)
Moderate renal dysfunction defined as GFR 30-60 ml/min/1.73m2 (Renal and urinary disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02561130/Prot_SAP_000.pdf